CLINICAL TRIAL: NCT07374497
Title: Effect of Perineal Massage on the Frequency of Episiotomy and Perineal Tearing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Principal Investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sheikh ZMC/H4
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Episiotomy Extended by Laceration
Keywords: Perineal massage; Vaginal delivery; Episiotomy; Perineal laceration; Perineal tear; Obstetric perineal injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapartum Perineal Massage Group (Experimental): Women received routine intrapartum care plus standardized intrapartum perineal massage performed by a trained doctor during the first stage of labour (repeated sessions) and an additional session as the second stage approached, using a sterile water-based obstetric lubricant.
  Interventions: Procedure: Intrapartum perineal massage
- Control Group (Placebo Comparator): Standard Intrapartum Care
  Interventions: Other: Standard Intrapartum Care Group (Control)

INTERVENTIONS:
Procedure: Intrapartum perineal massage — Standardized technique with gloved hands and water-based lubricant; thumbs introduced ~2-3 cm into the vagina with steady lateral pressure to vaginal side walls during resting intervals, delivered as 10-minute sessions repeated during first stage of labour, with an additional session near second stage; discontinued if bleeding, severe pain, suspected infection, non-reassuring fetal status, or urgent obstetric indication arose.
  Arms: Intrapartum Perineal Massage Group
Other: Standard Intrapartum Care Group (Control) — Women received routine intrapartum care only, with no perineal stretching or massage manoeuvres beyond routine perineal support during delivery, as per hospital protocols.
  Arms: Control Group

SUMMARY:
A randomized controlled trial was conducted at the Department of Obstetrics and Gynaecology, Sheikh Zayed Hospital, Rahim Yar Khan, over 6 months following Institutional Review Board and College of Physicians and Surgeons Pakistan approval, to assess whether intrapartum perineal massage reduces mediolateral episiotomy and lowers the frequency and severity of perineal tears in women undergoing term (37-42 weeks), singleton, cephalic vaginal delivery. Women aged 18-45 years in active labour who provided written informed consent were consecutively enrolled and randomized (1:1) by a computer-generated sequence with sequentially numbered, opaque, sealed envelopes to either standard intrapartum care or standard care plus perineal massage; women with conditions requiring urgent delivery/caesarean section or contraindicating vaginal delivery/perineal manipulation were excluded. In the intervention arm, a trained doctor performed standardized perineal massage using sterile water-based lubricant during the first stage and again near the second stage, with predefined stopping criteria for safety; the control arm received routine care without massage beyond usual perineal support at delivery. Primary outcomes were episiotomy (Yes/No) and perineal tear occurrence and grade (first-fourth), assessed immediately post-delivery by a consultant obstetrician not involved in providing massage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years
* Primigravida and multigravida women in active labor.
* Singleton, cephalic presentation of the fetus.
* Women who provide informed consent to participate in the study.
* Women at Term pregnancy (37 - 42 weeks).

Exclusion Criteria:

* Women with placental abruption, vaginal bleeding, macrosomia, fetal distress, vaginal infections, placenta previa and preterm births.
* Non-vertex fetal presentations such as breech.
* Women scheduled for a cesarean section.
* Pregnancies with multiple gestations (e.g., twins, triplets).
* Presence of active genital herpes or other contraindications to vaginal birth (HIV).
* Active vaginal infections, including bacterial vaginosis or yeast infections.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 202 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of episiotomy | Immediately at the time of delivery (during second stage and recorded immediately after birth)
  Proportion of participants in whom a mediolateral episiotomy was performed during vaginal delivery, based on predefined clinical indications and documented by the consultant obstetrician.
Frequency of perineal tears | Immediately after birth (post-delivery examination in the labour room)
  Proportion of participants with any spontaneous perineal laceration after vaginal delivery, determined on systematic post-delivery perineal and vaginal examination by the consultant obstetrician.

CONTACTS AND LOCATIONS:
Overall Officials: Sumbal Amjad, Principal Investigator — Sheikh Zayed Medical college/Hospital, Rahimyar Khan
Locations (1):
- Sheikh Zayed Medical college/hospital, Rahim Yar Khan, Punjab Province, Pakistan